CLINICAL TRIAL: NCT06579157
Title: The Association Between Pressure-Sensing Mattresses and Mechanical Ventilation Weaning in Neonatal
Brief Title: Pressure-Sensing Mattresses and Mechanical Ventilation Weaning in Neonatal
Status: Recruiting | Type: Observational
Sponsor: Fu Jen Catholic University (Other)
Responsible Party: Principal Investigator, Ke-Yun, Chao, Group leader of Respiratory Therapists, Fu Jen Catholic University
Other Study IDs: FJUH113387
Record Dates: First submitted 2024-08-27; First posted 2024-08-30 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: newborn; ballistocardiograph; pressure sensor; unobtrusive sensing
MeSH Terms: conditions — Bronchopulmonary Dysplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Pressure-Sensing Mattresses — using ballistocardiography (BCG) for monitoring respiration and heart rate in neonates

SUMMARY:
This study aims to explore the correlation between using ballistocardiography for monitoring respiration and heart rate in neonates under invasive and non-invasive respiratory support.

DETAILED DESCRIPTION:
Background： Traditional physiological measurement methods often require subjects to remain immobile or have various devices attached to their bodies, causing discomfort, especially unsuitable for neonatal care. However, with the development of electronic technologies, these methods have improved. ballistocardiography (BCG) presents a possible solution for monitoring neonates' physiological signals. BCG is a non-invasive and non-contact instrument that measures the body's reactive motion pressure changes caused by cardiac contraction. These sensors do not require direct attachment, allowing for long-term physiological signal measurement without disturbing the subject.

Methods： The study will be conducted in the neonatal intensive care unit on the seventh floor of Fu Jen Catholic University Hospital, with an expected enrollment of 60 participants. The subjects will be grouped and stratified based on weight and the use of invasive respiratory support. During the hospitalization, daily output of ventilator data and physiological monitor data will be collected and analyzed for correlation.

Effect： This trial is expected to confirm the application of BCG in the neonatal population, demonstrate its correlation with current conventional physiological monitors, and assess its applicability in low-weight preterm infants. Additionally, the study will investigate whether continuous BCG monitoring during hospitalization can predict the possibility of bronchopulmonary dysplasia.

ELIGIBILITY:
Inclusion Criteria:

* Using invasive ventilation support with flow sensors or non-invasive ventilation support
* The legal representative signs the informed consent form

Exclusion Criteria:

* Refusal to participate in the study

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: infant of Affiliated University Hospital
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-11-10 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
ballistocardiography waveform | through study completion, an average of 2 weeks
  the correlation between using Ballistocardiography (BCG) for monitoring respiration and heart rate

SECONDARY OUTCOMES:
tidal volume | through study completion, an average of 2 weeks
  the correlation between using Ballistocardiography (BCG) for tidal volume

CONTACTS AND LOCATIONS:
Overall Officials: Ke-Yun Chao, PhD, Principal Investigator — Fu Jen Catholic University Hospital
Locations (1):
- Fu Jen Catholic University Hospital, Fu Jen Catholic University, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No